CLINICAL TRIAL: NCT00275210
Title: Multicenter International Study of Oxaliplatin/ 5FU-LV in the Adjuvant Treatment of Colon Cancer
Brief Title: MOSAIC - Multicenter International Study of Oxaliplatin/ 5FU-LV in the Adjuvant Treatment of Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC3313
Record Dates: First submitted 2006-01-03; First posted 2006-01-11 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Colonic Neoplasms
Keywords: Oxaliplatin; Chemotherapy,adjuvant; Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin (SR96669)

SUMMARY:
To evaluate the FOLFOX regimen versus LV5FU2 in the adjuvant treatment of stage II and III colon cancer.

Primary objective: Disease Free Survival (DFS) Secondary objective: Overall Survival (OS), safety (including long term toxicity)

ELIGIBILITY:
Main selection criteria:

* Histologically proven stage Dukes " B2 " (stage II: T3-T4 N0 M0) and " C " (stage III: any T N1-2 M0) colon carcinoma. The inferior pole of the tumor must be above the peritoneal reflection (> 15 cm from the anal margin)·
* Complete resection of the primary tumor without gross or microscopic evidence of residual disease
* Treatment within 7 weeks following surgery
* Age 18-75 years old
* ECOG PS £ 2
* No prior chemo, immuno or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2246 (Actual)
Dates: Start 1998-10; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To to detect occurrence of relapse the following examinations have to be performed for 5 years:
Every 6 months for ultrasound or abdominopelvic CT scan and CEA determination,
Every year for chest X-ray and colonoscopy for non polyp free patient,
Every 3 years colonoscopy for polyp free patient

SECONDARY OUTCOMES:
Every 2 weeks clinical and laboratory tests (hematological, creatinine and liver tests) for safety evaluation during treatment then every 6 months neurological examination Date of death for OS

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, MD, Study Chair — Hopital saint-Antoine, Oncology department
Locations (19):
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Webster-Clark M, Keil AP, Robert N, Frytak JR, Boyd M, Sturmer T, Sanoff H, Westreich D, Lund JL. Comparing Trial and Real-world Adjuvant Oxaliplatin Delivery in Patients With Stage III Colon Cancer Using a Longitudinal Cumulative Dose. JAMA Oncol. 2022 Oct 13;8(12):1821-4. doi: 10.1001/jamaoncol.2022.4445. Online ahead of print. PMID 36227604
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Salem ME, Yin J, Goldberg RM, Pederson LD, Wolmark N, Alberts SR, Taieb J, Marshall JL, Lonardi S, Yoshino T, Kerr RS, Yothers G, Grothey A, Andre T, De Gramont A, Shi Q. Evaluation of the change of outcomes over a 10-year period in patients with stage III colon cancer: pooled analysis of 6501 patients treated with fluorouracil, leucovorin, and oxaliplatin in the ACCENT database. Ann Oncol. 2020 Apr;31(4):480-486. doi: 10.1016/j.annonc.2019.12.007. Epub 2020 Jan 16. PMID 32085892
- [Derived] Auclin E, Andre T, Taieb J, Banzi M, Van Laethem JL, Tabernero J, Hickish T, de Gramont A, Vernerey D. Association of post-operative CEA with survival and oxaliplatin benefit in patients with stage II colon cancer: a post hoc analysis of the MOSAIC trial. Br J Cancer. 2019 Aug;121(4):312-317. doi: 10.1038/s41416-019-0521-7. Epub 2019 Jul 12. PMID 31296923
- [Derived] Andre T, de Gramont A, Vernerey D, Chibaudel B, Bonnetain F, Tijeras-Raballand A, Scriva A, Hickish T, Tabernero J, Van Laethem JL, Banzi M, Maartense E, Shmueli E, Carlsson GU, Scheithauer W, Papamichael D, Moehler M, Landolfi S, Demetter P, Colote S, Tournigand C, Louvet C, Duval A, Flejou JF, de Gramont A. Adjuvant Fluorouracil, Leucovorin, and Oxaliplatin in Stage II to III Colon Cancer: Updated 10-Year Survival and Outcomes According to BRAF Mutation and Mismatch Repair Status of the MOSAIC Study. J Clin Oncol. 2015 Dec 10;33(35):4176-87. doi: 10.1200/JCO.2015.63.4238. Epub 2015 Nov 2. PMID 26527776
- [Derived] Tournigand C, Andre T, Bonnetain F, Chibaudel B, Lledo G, Hickish T, Tabernero J, Boni C, Bachet JB, Teixeira L, de Gramont A. Adjuvant therapy with fluorouracil and oxaliplatin in stage II and elderly patients (between ages 70 and 75 years) with colon cancer: subgroup analyses of the Multicenter International Study of Oxaliplatin, Fluorouracil, and Leucovorin in the Adjuvant Treatment of Colon Cancer trial. J Clin Oncol. 2012 Sep 20;30(27):3353-60. doi: 10.1200/JCO.2012.42.5645. Epub 2012 Aug 20. PMID 22915656